CLINICAL TRIAL: NCT07179068
Title: Protocol for a Pilot Randomized Trial Assessing the Acceptability, Feasibility, and Initial Efficacy of a Single-session Online Parent-focused Intervention Targeting Predictors of Body Image Disturbance in Young Children
Brief Title: Acceptability and Feasibility of a Single-Session Online Parent-Focused Intervention Targeting Child Body Image Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University at Albany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PrBI1243; 24-0041UA (Other Grant/Funding Number: The Caplan Foundation for early childhood)
Record Dates: First submitted 2025-08-26; First posted 2025-09-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Eating Disorders; Body Image Disturbance; Weight Bias
Keywords: Eating Disorder Prevention; Restriction; Loss of Control Eating; Body Image; Single Session Intervention
MeSH Terms: conditions — Feeding and Eating Disorders; Weight Prejudice

STUDY DESIGN:
Intervention Model Description: For the initial phase of the study, investigators will randomize 24 participants to one of the four modules in the study and receive detailed qualitative feedback from those participants (6 assigned to each module; 3 mothers and 3 fathers). For the second phase of the study (the randomized controlled trial portion of the project), which assesses acceptability, feasibility, and initial efficacy, investigators will randomize 100 parents to either the intervention group or the control group. The intervention group will view the entire intervention (all 4 modules) and complete knowledge checks at the end of the intervention. The control group will only complete the knowledge checks. Investigators will compare performance on the knowledge checks in the treatment and control groups as a measure of initial efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In phase 2, 50 participants will be randomized to complete the entire intervention; the intervention/workshop will consist of four modules: Body Image Development/Body Talk, Food Talk, Picky Eating and Mealtime Conversations, and Media Usage and Social Comparison. Each module will be approximately 10 minutes. After parents complete all four modules, they will complete measures of acceptability and feasibility, including reporting which module they found most useful. They will also complete knowledge checks.
  Interventions: Behavioral: Child Body Image Development Workshop
- Control (No Intervention): In Phase 2, 50 parents will be randomized into the control group. This group will receive no intervention. They will only complete the knowledge checks. These knowledge checks will be the same checks completed by the intervention group.

INTERVENTIONS:
Behavioral: Child Body Image Development Workshop — This is an online, single-session, modular intervention for parents of children that are two-to-six years old. It is designed to target and improve child body image development by providing psychoeducation and interactive activities to parents in each of the four modules. Modules include Body Image Development/Body Talk, Food Talk, Picky Eating and Mealtime Conversations, and Media Usage and Social Comparison. These modules were designed using the results of our previously completed Needs Assessment, as well as the current evidence-base regarding risk factors for the development of body image in young children.
  Arms: Intervention

SUMMARY:
Body image concerns have been linked to diverse mental health issues, including depression and disordered eating. Disordered eating can develop into clinically significant eating disorders, which are associated with serious negative impacts on psychological and physical well-being, and can adversely impact developmental trajectories in children and adolescents. Given limitations in the eating disorder intervention literature, it is important to invest in effective eating disorder prevention programs. Evidence suggests that children can recognize the existence of societal appearance ideals as early as age 3; thus, this study examines the acceptability and feasibility of a single-session, online, parent-focused intervention targeting predictors of body image disturbance in young children.

DETAILED DESCRIPTION:
Body image concerns have been linked longitudinally to diverse mental health issues, including disordered eating. Disordered eating can develop into clinically significant eating disorders, which are associated with serious psychological and physical sequelae and can adversely impact developmental trajectories in children and adolescents. The mortality rate associated with eating disorders is second only to that of opiate addiction. Existing treatments for eating disorders remain only moderately effective, with ~40% remission rates for anorexia and bulimia nervosa. It is therefore important to examine early risk factors for the development of body image concerns to inform preventive approaches suitable for intervening early on in the development of disordered eating.

Evidence suggests that children can recognize the existence of societal appearance ideals as early as age 3; in fact, exposure to appearance-focused media at age 3 is prospectively predictive of positive associations with thinness at age 4 and dietary restraint behaviors at age 5. These findings suggest an important role of societal appearance ideals in fostering body discontent and point to the media as a crucial source of communication of these ideals to children. Parents have a great deal, if not all, control over the information their young children are exposed to within the home and from the outside world. The proposed study is based on the assumption that intervening with parents of young children, with a focus on education about the impact of media exposure, can reduce body image disturbance and prevent the future development of disordered eating. Thus, this study explores the acceptability and feasibility of a single-session, online, parent-focused intervention targeting predictors of body image disturbance in young children.

ELIGIBILITY:
Inclusion Criteria: Must be at least 18 years old and reside in the US. They must also be the parent of a young child between the ages of 2-6.

Exclusion Criteria: None beyond not meeting inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Investigators will recruit an equal number of mothers and fathers. In Phase 1, investigators will recruit 12 mothers and 12 fathers. In Phase 2, investigators will recruit 50 mothers and 50 fathers.
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Directly after completion of the intervention.
  Acceptability will be examined via questions about intervention credibility and expectancy to be completed by workshop participants post-intervention, adapted from the well-establish Credibility and Expectancy Questionnaire (e.g., "At this point, how logical does the intervention seem to you?" "At this point, how successful do you think this information will be in reducing your concerns about your child's eating patterns?").
Recruitment | 1 year after study recruitment begins.
  Feasibility includes recruitment and retention rates and measurement burden. First, feasibility will be defined as successful recruitment of 50 moms and 50 dads.
Retention | At the end of data collection, an average of one year after recruitment begins.
  Feasibility includes recruitment and retention rates and measurement burden. Second, feasibility will be defined as retention of 85 % of participants through the entire intervention.
Missingness | At the end of data collection, an average of one year after recruitment begins.
  In addition, minimal missing data as well as survey items completed will be looked at as measures of feasibility. Less than 5 % of missing data will be required for the study to be considered feasible.

SECONDARY OUTCOMES:
Initial Efficacy | Directly following completion of the intervention.
  In Phase 2, 50 parents in the intervention group will complete the intervention, and then complete knowledge checks. 50 parents in the control group will not complete the intervention, and will only complete the knowledge checks. As a measure of initial efficacy, a t-test will be used to compare performance on the knowledge checks in the treatment vs. control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Prolific Online Survey Platform, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No